CLINICAL TRIAL: NCT03517267
Title: Validation of the New Thyroid Imaging Reporting and Data System (TIRADS) From 2017 Risk Assessment of Thyroid Nodules in Comparison to the American Thyroid Association (ATA) Guidelines From 2015
Brief Title: Thyroid Imaging Reporting and Data System (TIRADS ) Versus Thyroid Association (ATA) Guidelines
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, razi-Beck Nira MD, Director Ultrasound Unit, Rambam Health Care Campus
Other Study IDs: : RambamMC
Record Dates: First submitted 2018-03-28; First posted 2018-05-07 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound and FNA — The nodule to undergo FNA will be chosen according to TIRADS ACR criteria and the ATA risk criteria ( if there is a disagreement between the methods whether to perform FNA the FNA will be performed ) If both methods do not recommend FNA , but the referring doctor has requested the procedure or the patient is unable to stay on follow up , the FNA will be performed .

SUMMARY:
Thyroid nodules are a very common clinical problem with prevalence of up to 68% in adults on high-resolution ultrasound .Ultrasound used in order to differentiate between benign and malignant lesion in the thyroid has shown sensitivity of 93.8% and specificity of 66% and US guided ( Fine needle aspiration ) FNA is known to be the test of choice in order to determine the nodules nature . Four to 6.5 % of all nodules are malignant .There are several guidelines that were suggested to help predict the risk stratification of thyroid nodules by ultrasound .

The American Thyroid Association (ATA) is widely used as evaluation, clinical and ultrasound criteria for fine-needle aspiration biopsy and management of thyroid nodules. The recent ACR TIRADS is a reporting system for thyroid nodules on ultrasound proposed by the American College of Radiology (ACR) published april 2017 that uses a slightly different scoring system for recommendation for FNA of thyroid.

The aim of this study is to validate TIRADS ACR 2017 risk stratification in the patient population in comparison to ATA risk stratification

DETAILED DESCRIPTION:
Thyroid nodules are a very common clinical problem with prevalence of up to 68% in adults on high-resolution ultrasound .Ultrasound used in order to differentiate between benign and malignant lesion in the thyroid has shown sensitivity of 93.8% and specificity of 66% and US guided ( Fine needle aspiration ) FNA is known to be the test of choice with sensitivity and specificity were 89.5% and 98%, respectively in order to determine the nodules nature, . Four to 6.5 % of all nodules are malignant .There are several guidelines that were suggested to help predict the risk stratification of thyroid nodules by ultrasound .

The American Thyroid Association (ATA) guidelines which characterized the nodule by its size, echogenicity, shape, presence or absence of calcification and evidence of Extrathyroidal extension (ETE) is widely use as evaluation, clinical and ultrasound criteria for fine-needle aspiration biopsy and management of thyroid nodules. These nodule characteristics classify the risk for malignancy into five categories which include benign pattern, very low suspicion pattern, low suspicion pattern, intermediate suspicious pattern and high suspicion pattern .

The recent ACR TIRADS is a reporting system for thyroid nodules on ultrasound proposed by the American College of Radiology (ACR) published april 2017 that uses a slightly different scoring system for recommendation for FNA of thyroid nodules .The ultrasound features set by TIRADS include composition, echogenicity, shape, margins and echogenic foci. The scoring range according suspicion of malignancy.

The aim of this study is to validate TIRADS ACR 2017 risk stratification in the patient population in comparison to ATA risk stratification.

Methods

The study will be prospective Informed consent will be signed before the FNA All patients referred for thyroid nodule FNA from outpatient and in patient clinics over 18 will be included .

The nodule to undergo FNA will be chosen according to TIRADS ACR criteria and the ATA risk criteria ( if there is a disagreement between the methods whether to perform FNA the FNA will be performed ) If both methods do not recommend FNA , but the referring doctor has requested the procedure or the patient is unable to stay on follow up , the FNA will be performed .

Data will be collected according the table Cytological results using Bethesda scoring and surgery results, when applicable will be collected .

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for thyroid nodule FNA from outpatient and in patient clinics
* Patients older that 18

Exclusion Criteria:

# Patients younger that 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred for thyroid nodule FNA
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Validation of Risk stratifications | The outcome measures will be assessed within 1 year from the initiation of recruitment.
  All nodules that will be aspirated , will be categorized according to the two risk stratification methods:
  Thyroid Imaging Reporting and Data System (TIRADS) and the American Thyroid Association (ATA) guidelines. The cytology results will be documented in the form of Bethesda scoring The risk stratification results will be compared to the Cytology results that will be considered the gold standard for malignancy .
  Accuracy of each method will be calculated .

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israek, Israel

IPD SHARING:
Plan to Share IPD: No